CLINICAL TRIAL: NCT04432493
Title: Using Combined EEG and Non-invasive Brain Stimulation to Examine and Improve Reward Functioning in Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Travis Baker, PhD, Principal Investigator, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2018002739
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Opioid-use Disorder
Keywords: Transcranial magnetic stimulation; Reward processing; Cognitive control
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded as to TMS condition (active or sham)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active TMS - OUD (Experimental): Participants in the opioid used disorder group (OUD) in the active condition will receive repetitive TMS (rTMS), delivered at 110% of participants' resting motor threshold at 10 Hz continuously over the predefined DLFPC target for a total of 2000 pulses
  Interventions: Device: Active repetitive transcranial magnetic stimulation (rTMS)
- Sham TMS - OUD (Placebo Comparator): Identical parameters will be applied to the opioid used disorder (OUD) SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation
  Interventions: Device: Sham repetitive transcranial magnetic stimulation (rTMS)
- Active TMS - HC (Active Comparator): Healthy Control (HC) participants in the active condition will receive repetitive TMS (rTMS), delivered at 110% of participants' resting motor threshold at 10 Hz continuously over the predefined DLFPC target for a total of 2000 pulses
  Interventions: Device: Active repetitive transcranial magnetic stimulation (rTMS)
- Sham TMS - HC (Sham Comparator): Identical parameters will be applied to the healthy control (HC) SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation
  Interventions: Device: Sham repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Active repetitive transcranial magnetic stimulation (rTMS) — rTMS will be used to stimulate neuronal activity of the dorsolateral prefrontal cortex (DLPFC). Participants will receive no more than 2000 pulses of rTMS at 110% of participants' resting motor threshold at 10 Hz continuously for the duration of the t-maze task.
  Arms: Active TMS - HC; Active TMS - OUD
Device: Sham repetitive transcranial magnetic stimulation (rTMS) — Sham TMS will be used to mimic the auditory sensation of the Active rTMS condition. Protocols for the sham condition will be the same as the active condition, however the TMS coil will be flipped 180 degrees so that participants in this condition will not receive any active stimulation.
  Arms: Sham TMS - HC; Sham TMS - OUD

SUMMARY:
The primary aims of this study are to identify impaired cognitive control in opioid use disorder (OUD) and subsequently to examine the effects of transcranial magnetic stimulation (TMS) on reward processing, as measured by the reward positivity (an electrophysiological signal) in people with OUD. To this end, the investigators will adopt a randomized sham-controlled trial to evaluate the efficacy of Ri-TMS on cognitive control in OUD.

The investigators hypothesize that Ri-TMS will be successful in modulating the reward positivity in opioid users in the active TMS condition.

DETAILED DESCRIPTION:
The design is primarily a randomized control-trial design, comparing the effects of placebo (sham) and active TMS stimulation on reward processing across two groups of participants - healthy controls and opioid users.

Participants will be asked to engage in a virtual T-maze task, a reward-based choice task that elicits robust reward positivities. During this task participants will receive simultaneous EEG/TMS, while they engage in the virtual T-maze decision making task, used in our previous reward positivity studies on SUDs. ERPs will be recorded throughout the T-Maze task, and the reward positivity will be measured as the difference in maximum amplitude between reward and no-reward feedback conditions.

The TMS coil will be positioned using a an Adept Viper s850 robotic arm (SmartMove, ANT Neuro, Enschede, The Netherlands), providing precise targeting of the predetermined left dorsolateral prefrontal (DLPFC) coordinate (< 10 mm from the scalp, orientated at a 45º angle). Participants in the active TMS condition will receive rTMS pulses throughout the duration of the T-Maze task, with a maximum of 2000 pulses delivered to each participant. Identical parameters will be applied to the SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Native English speakers
* Males and Females aged 18-55 years old
* Ability to provide informed written or verbal consent
* Opioid dependent individuals (according to the Alcohol, Smoking and Substance Involvement Screening Test opioid dependence score), or
* Healthy controls with no history of significant substance use

Exclusion Criteria:

* Un-correctable visual impairment
* Uninterruptable central nervous system medication
* TMS contraindications (e.g., pregnancy, braces, history of seizures, metal implants).
* History of neurological or psychiatric illness
* Diagnosed learning disability
* History of significant head injury (loss of consciousness for more than five minutes)
* Substance abuse (Participants who score above 39.5 on the Global Continuum of Substance Risk scale of the Alcohol, Smoking and Substance Involvement Screening Test - controls only)
* Use of psychoactive or vasoactive medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Biernacki, PhD, Principal Investigator — Rutgers University - Newark
Locations (1):
- Rutgers University - Newark, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Data may be uploaded to an open source framework. All data will be de-identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TMS - OUD: OUD Participants in the active condition will receive repetitive TMS (rTMS), delivered at 110% of participants' resting motor threshold at 10 Hz continuously over the predefined DLFPC target for a total of 2000 pulses
  Active repetitive transcranial magnetic stimulation (rTMS): rTMS will be used to stimulate neuronal activity of the dorsolateral prefrontal cortex (DLPFC). Participants will receive no more than 2000 pulses of rTMS at 110% of participants' resting motor threshold at 10 Hz continuously for the duration of the t-maze task.
- Sham TMS - OUD: Identical parameters will be applied to the OUD SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation
  Sham repetitive transcranial magnetic stimulation (rTMS): Sham TMS will be used to mimic the auditory sensation of the Active rTMS condition. Protocols for the sham condition will be the same as the active condition, however the TMS coil will be flipped 180 degrees so that participants in this condition will not receive any active stimulation.
- Active TMS - HC: Health Control (HC) Participants in the active condition will receive repetitive TMS (rTMS), delivered at 110% of participants' resting motor threshold at 10 Hz continuously over the predefined DLFPC target for a total of 2000 pulses Active repetitive transcranial magnetic stimulation (rTMS): rTMS will be used to stimulate neuronal activity of the dorsolateral prefrontal cortex (DLPFC). Participants will receive no more than 2000 pulses of rTMS at 110% of participants' resting motor threshold at 10 Hz continuously for the duration of the t-maze task.
- Sham TMS - HC: Identical parameters will be applied to the healthy control (HC) SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation Sham repetitive transcranial magnetic stimulation (rTMS): Sham TMS will be used to mimic the auditory sensation of the Active rTMS condition. Protocols for the sham condition will be the same as the active condition, however the TMS coil will be flipped 180 degrees so that participants in this condition will not receive any active stimulation.
Period: Overall Study
Arm/Group | Active TMS - OUD | Sham TMS - OUD | Active TMS - HC | Sham TMS - HC
Started | 16 | 18 | 22 | 25
Completed | 16 | 18 | 22 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active TMS - OUD: Opioid Use Disorder (OUD) Participants in the active condition will receive repetitive TMS (rTMS), delivered at 110% of participants' resting motor threshold at 10 Hz continuously over the predefined DLFPC target for a total of 2000 pulses
  Active repetitive transcranial magnetic stimulation (rTMS): rTMS will be used to stimulate neuronal activity of the dorsolateral prefrontal cortex (DLPFC). Participants will receive no more than 2000 pulses of rTMS at 110% of participants' resting motor threshold at 10 Hz continuously for the duration of the t-maze task.
- Sham TMS - OUD: Identical parameters will be applied to the Opioid Use Disorder (OUD) SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation
  Sham repetitive transcranial magnetic stimulation (rTMS): Sham TMS will be used to mimic the auditory sensation of the Active rTMS condition. Protocols for the sham condition will be the same as the active condition, however the TMS coil will be flipped 180 degrees so that participants in this condition will not receive any active stimulation.
- Total: Total of all reporting groups
Arm/Group | Active TMS - OUD | Sham TMS - OUD | Active TMS - HC | Sham TMS - HC | Total
Number analyzed (Participants) | 16 | 18 | 22 | 25 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 22 | 25 | 81
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (9) | 46 (19) | 36 (12) | 34 (11) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 10 | 12 | 33
  Male | 11 | 12 | 12 | 13 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 12 | 10 | 8 | 40
  White | 4 | 6 | 7 | 11 | 28
  More than one race | 1 | 0 | 3 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: μV (Microvolts]
  United States | 16 | 18 | 22 | 25 | 81

OUTCOME MEASURES:

1. Primary Outcome: Reward Positivity
Description: The reward positivity is an event-related brain potential, sensitive to reward feedback. The reward positivity will be measured during the t-maze task, where participants will receive feedback on choices (Reward, No-reward). Reward positivity amplitude will be determined by identifying the maximum absolute amplitude of the difference wave within a 200- to 400-ms window following feedback onset. The reward positivity will be evaluated along front-central electrodes (Fz, FCz, Cz).
Time Frame: Day 0 (day of testing)
Measure: Mean (Standard Deviation); unit: μV (microvolts)
Groups:
- Active TMS - OUD; Active TMS - Controls; Sham TMS - Controls: Participants in the active condition will receive repetitive TMS (rTMS), delivered at 110% of participants' resting motor threshold at 10 Hz continuously over the predefined DLFPC target for a total of 2000 pulses
  Active repetitive transcranial magnetic stimulation (rTMS): rTMS will be used to stimulate neuronal activity of the dorsolateral prefrontal cortex (DLPFC). Participants will receive no more than 2000 pulses of rTMS at 110% of participants' resting motor threshold at 10 Hz continuously for the duration of the t-maze task.
- Sham TMS - OUD: Identical parameters will be applied to the SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation
  Sham repetitive transcranial magnetic stimulation (rTMS): Sham TMS will be used to mimic the auditory sensation of the Active rTMS condition. Protocols for the sham condition will be the same as the active condition, however the TMS coil will be flipped 180 degrees so that participants in this condition will not receive any active stimulation.
Arm/Group | Active TMS - OUD | Sham TMS - OUD | Active TMS - Controls | Sham TMS - Controls
Number analyzed (Participants) | 16 | 18 | 22 | 24
μV (microvolts) | -5.2 (2) | -2.3 (3) | -4.4 (3) | -4.6 (3)

ADVERSE EVENTS:
Time Frame: through study completion (e.g. on the day of testing).
Arm/Group | Active TMS - OUD | Sham TMS - OUD | Active TMS - Controls | Sham TMS - Controls
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18 | 0/22 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/22 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT04432493/Prot_003.pdf
  • Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT04432493/SAP_004.pdf
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT04432493/ICF_005.pdf